CLINICAL TRIAL: NCT02335294
Title: A Phase 2, Randomized, Double-Blind, Placebo- and Active-controlled Study of TRV130 for the Treatment of Acute Postoperative Pain Following Abdominoplasty
Brief Title: A Study of TRV130 for the Treatment of Pain After Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP130-2002
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: Pain; abdominoplasty; PCA
MeSH Terms: conditions — Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TRV130 (Experimental)
  Interventions: Drug: TRV130
- Morphine (Active Comparator)
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRV130 — Rescue: Ibuprofen, oxycodone
  Arms: TRV130
Drug: Morphine — Rescue: Ibuprofen, oxycodone
  Other Names: Morphine sulphate
  Arms: Morphine
Drug: Placebo — Rescue: Ibuprofen, oxycodone
  Other Names: Dextrose 5% in water, D5W
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of IV TRV130 compared with placebo in patients with acute postoperative pain following abdominoplasty.

DETAILED DESCRIPTION:
The primary objective is to evaluate the analgesic efficacy of intravenous (IV) TRV130 administered via patient controlled analgesia device (PCA) compared with placebo administered via PCA in patients with moderate to severe, acute postoperative pain following abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* >=18 and <=65 years of age.
* Plans to undergo an abdominoplasty procedure with no additional collateral procedures.
* Is able to understand and comply with the procedures and study requirements, and to provide written informed consent before any study procedure.

Exclusion Criteria:

* ASA Physical Status Classification System classification of P3 or worse.
* Has surgical or post-surgical complications.
* Has clinically significant medical conditions or history of such conditions that may interfere with the interpretation of efficacy, safety, or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Has previously participated in another TRV130 clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pasadena, California
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Protocol v1-4 TRV130 0.1 mg: TRV130 loading doses totaling 1.5 mg. TRV130 0.1 mg PCA with 6-min lockout.
- Protocol v1-4 Morphine; Protocol v5 Morphine: Morphine loading doses totaling 4 mg. Morphine 1 mg PCA with 6-min lockout.
- Protocol v1-4 Placebo; Protocol v5 Placebo: Placebo (5% D5W) loading doses totaling 4 ml. Placebo 1 ml PCA with 6-min lockout.
- Protocol v5 TRV130 0.35 mg: TRV130 loading doses totaling 1.5 mg. TRV130 0.35 mg PCA with 6-min lockout.
Period: Overall Study
Arm/Group | Protocol v1-4 TRV130 0.1 mg | Protocol v1-4 Morphine | Protocol v1-4 Placebo | Protocol v5 TRV130 0.35 mg | Protocol v5 Morphine | Protocol v5 Placebo
Started | 39 | 42 | 19 | 39 | 41 | 20
Completed | 36 | 38 | 18 | 36 | 39 | 19
Not Completed | 3 | 4 | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocol v1-4 TRV130 0.1 mg | Protocol v1-4 Morphine | Protocol v1-4 Placebo | Protocol v5 TRV130 0.35 mg | Protocol v5 Morphine | Protocol v5 Placebo | Total
Number analyzed (Participants) | 39 | 42 | 19 | 39 | 41 | 20 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 42 | 19 | 39 | 41 | 20 | 200
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.07) | 37.0 (9.23) | 36.6 (8.60) | 40.3 (11.987) | 38.4 (9.064) | 38.5 (10.018) | 38.2 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 19 | 39 | 41 | 18 | 198
  Male | 0 | 0 | 0 | 0 | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 5 | 16 | 16 | 5 | 71
  Not Hispanic or Latino | 24 | 28 | 14 | 23 | 25 | 15 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Asian | 0 | 2 | 0 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 2 | 0 | 0 | 3
  Black or African American | 12 | 15 | 10 | 18 | 17 | 10 | 82
  White | 27 | 24 | 8 | 18 | 21 | 9 | 107
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 19 | 39 | 41 | 20 | 200

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average (TWA) Change From Baseline in Pain Score Over 24 Hours Between TRV130 and Placebo
Description: Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 24 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (24 hours) to yield values on the 0-10 NPRS.
Time Frame: 24-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol v1-4 TRV130 0.1 mg | Protocol v1-4 Placebo | Protocol v5 TRV130 0.35 mg | Protocol v5 Placebo
Number analyzed (Participants) | 39 | 19 | 39 | 20
score on a scale | -3.8 (2.53) | -1.7 (2.26) | -3.5 (2.32) | -1.2 (2.93)

2. Secondary Outcome: Time Weighted Average (TWA) Change From Baseline in Pain Score Over 24 Hours Between TRV130 and Morphine
Description: as for outcome 1
Time Frame: 24-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol v1-4 TRV130 0.1 mg | Protocol v1-4 Morphine | Protocol v5 TRV130 0.35 mg | Protocol v5 Morphine
Number analyzed (Participants) | 39 | 42 | 39 | 41
score on a scale | -3.8 (2.53) | -3.4 (2.74) | -3.5 (2.32) | -3.6 (2.61)

ADVERSE EVENTS:
Arm/Group | Protocol v1-4 TRV130 0.1 mg | Protocol v1-4 Morphine | Protocol v1-4 Placebo | Protocol v5 TRV130 0.35 mg | Protocol v5 Morphine | Protocol v5 Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42 | 0/19 | 0/39 | 0/41 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/42 | 0/19 | 0/39 | 1/41 | 0/20
Other Adverse Events (participants affected / at risk) | 26/39 | 39/42 | 8/19 | 32/39 | 39/41 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Protocol v1-4 TRV130 0.1 mg (N=39) | Protocol v1-4 Morphine (N=42) | Protocol v1-4 Placebo (N=19) | Protocol v5 TRV130 0.35 mg (N=39) | Protocol v5 Morphine (N=41) | Protocol v5 Placebo (N=20)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Protocol v1-4 TRV130 0.1 mg (N=39) | Protocol v1-4 Morphine (N=42) | Protocol v1-4 Placebo (N=19) | Protocol v5 TRV130 0.35 mg (N=39) | Protocol v5 Morphine (N=41) | Protocol v5 Placebo (N=20)
Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 16 | 34 | 3 | 18 | 26 | 4
Vomiting (Gastrointestinal disorders) | 6 | 17 | 2 | 6 | 18 | 1
Local Swelling (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 4 | 1
Headache (Nervous system disorders) | 6 | 6 | 0 | 6 | 8 | 5
Presyncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 7 | 0 | 2 | 3 | 0
Tension Headache (Nervous system disorders) | 1 | 4 | 2 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 0 | 12 | 23 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 1 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 6 | 4 | 1 | 3 | 3 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion Site Discomfort (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Infusion Site Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Infusion Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Postoperative Fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T-Wave Abnormal (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomina (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other